CLINICAL TRIAL: NCT04526886
Title: A Pragmatic, Single-Arm Clinical Trial of a Novel Dose Adjustment Algorithm for Preventing Cytopenia-Related Delays During FOLFOX Chemotherapy
Brief Title: Clinical Trial of a Novel Dose Adjustment Algorithm for Preventing Cytopenia-Related Delays During FOLFOX Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gabriel A. Brooks, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20125
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Gastric Cancer; Esophageal Cancer; Ampullary Cancer; Small Bowel Cancer; Appendix Cancer
Keywords: neutropenia; thrombocytopenia; FOLFOX; dose adjustment
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Appendiceal Neoplasms; Neutropenia; Thrombocytopenia | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): All patients in this single-arm study will be exposed to the experimental chemotherapy dose-adjustment algorithm.
  Interventions: Other: Algorithm for cytopenia-related delay and dose-reduction of mFOLFOX chemotherapy

INTERVENTIONS:
Other: Algorithm for cytopenia-related delay and dose-reduction of mFOLFOX chemotherapy — Chemotherapy dose-adjustment algorithm for FOLFOX chemotherapy

SUMMARY:
The study is testing an intervention of an investigator-developed chemotherapy dose adjustment algorithm. The primary objective of this study is to evaluate the effectiveness of the chemotherapy dose adjustment algorithm for reducing unplanned delays in patients receiving FOLFOX (5-fluorouracil, leucovorin, and oxaliplatin)-type chemotherapy, while maintaining acceptable chemotherapy dose-intensity.

DETAILED DESCRIPTION:
The study intervention will involve implementation of a clinical algorithm to guide chemotherapy dose reductions and treatment delays in patients with neutropenia and/or thrombocytopenia during treatment with FOLFOX-type regimens. The clinical algorithm was developed by the principal investigator, and the algorithm has been iteratively revised over time based on experiences from use in routine care.

Features of the dose adjustment algorithm that differ from criteria used in clinical trial protocols and routine care include:

* At presentation for cycle 2 and 3 - the algorithm employs proactive chemotherapy dose reductions, without treatment delay, in patients with mild cytopenias (absolute neutrophil count [ANC] 1000-1499/mm3 and/or platelet count 75,000-99,000/mm3). In usual care, mild cytopenias during early treatment cycles do not trigger a chemotherapy dose reduction, but these early cytopenia events often lead to more severe cytopenias and subsequent delays in later treatment cycles.
* At any cycle - the algorithm employs chemotherapy dose reductions without treatment delay in patients with moderate cytopenias (ANC 750-999/mm3 and/or platelet count 50,000-74,000/mm3). In usual care, moderate cytopenias trigger both a chemotherapy treatment delay AND a subsequent dose reduction, whereas the study algorithm will introduce a dose reduction without a treatment delay.

Decisions about dose modifications and delays for reasons other than neutropenia and/or thrombocytopenia will be made at the discretion of the treating clinician, as per standard-of-care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Diagnosis of adenocarcinoma of the gastrointestinal tract (to include cancers of the colorectum, stomach, esophagus, appendix, and small bowel)
* The treating oncologist's recommendation must be for six or more cycles of standard-dose mFOLFOX chemotherapy (with or without concurrent bevacizumab, cetuximab, panitumumab, or trastuzumab). Intent of treatment may be either curative or palliative in nature.
* Completion of day 1 of cycle 1 of standard-of-care FOLFOX chemotherapy

Exclusion Criteria:

* Prior receipt of systemic chemotherapy in the 12 months prior to day 1 of cycle 1 of mFOLFOX (other than radiation-sensitizing chemotherapy)
* History of baseline neutropenia; defined as neutrophil count <1500 in the 30 days preceding planned day 1 of cycle 1 of mFOLFOX
* History of baseline thrombocytopenia; defined as platelet count <100,000) in the 30 days preceding planned day 1 of cycle 1 of mFOLFOX
* Patients with a history of an uncorrected bleeding condition that would preclude safe use of the dose adjustment algorithm, in the judgement of the enrolling investigator
* Patients who have started a new prescription anticoagulant (e.g. warfarin, heparin derivatives, or direct oral anticoagulants) in the 14 days preceding day 1 of cycle 1 of mFOLFOX
* Patients who are unable to provide informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel A Brooks, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kogan LG, Davis SL, Brooks GA. Treatment delays during FOLFOX chemotherapy in patients with colorectal cancer: a multicenter retrospective analysis. J Gastrointest Oncol. 2019 Oct;10(5):841-846. doi: 10.21037/jgo.2019.07.03. PMID 31602321
- [Derived] Wright HN, Tosteson TD, Hourdequin KC, Ripple GH, Fuld AD, Dragnev KH, Amin M, Muralikrishnan S, McGrath EB, Stannard MG, Schofield LL, Lord-Halvorson S, Tosteson ANA, Brooks GA. A pragmatic, single-arm clinical trial of a dose modification algorithm for preventing cytopenia-related delays during FOLFOX chemotherapy. Support Care Cancer. 2025 Aug 8;33(9):769. doi: 10.1007/s00520-025-09784-0. PMID 40779182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Dartmouth Cancer Center from the Lebanon, NH, St. Johnsbury, VT, and Nashua, NH, clinic sites between September 14, 2020 and December 14, 2022.
Period: Overall Study
Arm/Group | Study Arm
Started | 52
Completed | 48
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Groups:
- Evaluable Subjects: All patients in this single-arm study will be exposed to the experimental chemotherapy dose-adjustment algorithm.
  Algorithm for cytopenia-related delay and dose-reduction of mFOLFOX chemotherapy: Chemotherapy dose-adjustment algorithm for FOLFOX chemotherapy
Arm/Group | Evaluable Subjects
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 26
Age, Continuous [Median (Full Range); unit: Years] | 66 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Unplanned Chemotherapy Treatment Delay
Description: Number of patients with any interruption of chemotherapy leading to a cycle length of >18 days that is not anticipated as of day 3 of the preceding treatment cycle.
Time Frame: Through day 1 of cycle 6 of FOLFOX chemotherapy (cycle length is 14 days)
Measure: Count of Participants; unit: Participants
Groups:
- Evaluable Participants: All study participants evaluable for the primary outcome
Arm/Group | Evaluable Participants
Number analyzed (Participants) | 48
Participants | 16

2. Secondary Outcome: Composite Safety Endpoint
Description: Number of patients meeting the composite endpoint of 1) febrile neutropenia (grade 3 or 4), 2) major bleeding with concurrent grade 3 thrombocytopenia (platelet count <50,000/mm3), 3) CTCAE grade 4 neutropenia (ANC <500/mm3), and/or 4) CTCAE grade 4 thrombocytopenia (platelet count <25,000/mm3)
Time Frame: Through day 1 of cycle 6 of FOLFOX chemotherapy (cycle length is 14 days)
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Participants: All participants enrolled in the study - includes participants who were not evaluable for the primary study outcome
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 52
Participants | 3

3. Secondary Outcome: Relative Dose Intensity of Chemotherapy
Description: Relative dose intensity (RDI) of chemotherapy. RDI is defined as (planned cumulative dose/cumulative administered dose)*(actual duration/planned duration). RDI will be calculated separately for each component of the FOLFOX regimen (5-FU bolus, 5-FU infusion, oxaliplatin).
Time Frame: Through day 1 of cycle 6 of FOLFOX chemotherapy (cycle length is 14 days)
Measure: Mean (Inter-Quartile Range); unit: Percentage
Groups:
- Participants Completing Six Cycles of FOLFOX: Participants completing six cycles of FOLFOX (evaluable population for relative dose intensity)
Arm/Group | Participants Completing Six Cycles of FOLFOX
Number analyzed (Participants) | 45
Percentage
  5-FU infusion | 0.913 [0.875 to 1.00]
  Oxaliplatin | 0.850 [0.789 to 0.968]
  5-FU bolus | 0.643 [0.455 to 0.917]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between the date of registration and the day 1 of the cycle 6 of FOLFOX chemotherapy (14-day planned cycle length).
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 1/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 4/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants (N=52)
Neutropenia, Grade 4 (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT04526886/Prot_SAP_000.pdf